CLINICAL TRIAL: NCT01261364
Title: The Evaluation of the Clinical Impact of the Antidepressant Pharmacogenomic Algorithm in an Outpatient Clinical Setting:A Randomized Double Blind Pilot Study
Brief Title: Pharmacogenetic-Directed Treatment for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assurex Health Inc. (Industry)
Collaborators: Pine Rest Christian Mental Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10002
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: GeneSight; Assurex; AssureRx
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual
- Pharmacogenetic guided treatment (Experimental)
  Interventions: Behavioral: GeneSightRx

INTERVENTIONS:
Behavioral: GeneSightRx — Multi-genetic pharmacogenomic panel
  Arms: Pharmacogenetic guided treatment
Behavioral: Treatment as usual — Treatment as usual
  Arms: Treatment as Usual

SUMMARY:
Determine if antidepressant treatment guided by pharmacogenetic algorithm and interpretive report improves outcomes when compared with standard treatment without the availability of genetic information.

DETAILED DESCRIPTION:
This study is designed to evaluate the clinical impact of pharmacogenetic (PGx)-directed treatment, as guided by interpretive, algorithmic report in the Pine Rest outpatient behavioral health clinics. The PGx algorithm utilized in this study is the foundation of a novel method of interpreting genetic testing results and reports them in a rapidly delivered format that provides enhanced guidance to psychiatrists in their selection of antidepressant medications

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (296.2, 296.3) or Depressive Disorder NOS (311.0) by a board certified psychiatrist.
* The patient is referred to the study by their treating psychiatrist or nurse practitioner who is approved by the study investigators to make subject referrals to the study.
* The patient is an outpatient and not in imminent need of inpatient hospitalization for medical or psychiatric reasons.
* Patient's baseline 17-Item Hamilton Depression (HAMD17) Rating score is >14.
* Provide a copy of a physical exam report performed within 6 months prior to study enrollment or undergo a physical exam by either their personal physician, a physician who is a subinvestigator on the study, or a study-contracted physician assistant in internal medicine.
* Undergo a medical history that includes a review of major organ systems by either their treating clinician, a subinvestigator physician, or a study-contracted physician assistant in internal medicine.
* The patient has signed the study informed consent form.

Exclusion Criteria:

* Serious medical illness (as ascertained via inclusion criteria 6 and 7, above).
* Diagnosis of a Bipolar Disorder.
* Diagnosis of Schizophrenia or Schizoaffective disorder.
* Evidence from history, baseline urine drug screen, and/or psychiatric interview of active abuse of alcohol and/or other drugs of abuse within 6 months prior to study enrollment. Patients who occasionally use marijuana may still be eligible if it is determined through psychiatric interview that the level of use does not qualify as abuse, dependence, or addiction. Patients testing positive for opioids or benzodiazepines are eligible if there is no evidence of abuse and it is determined that they are taking opioid analgesics or a benzodiazepine that is prescribed by a licensed prescriber for a medical or psychiatric indication.
* History of prior pharmacogenomic testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Depression Score reduction | 8 weeks
  Mean change in the 17 item Grid Hamilton Depression (HAMD17) score from baseline at each assessment.
Side effect reduction | 8 weeks
  Mean change in the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) score from baseline at each assessment.

SECONDARY OUTCOMES:
Depression response or remission | 8 weeks
  Percentage of subjects who respond (≥50% decrease in HAMD17 and QIDS-CR* rating) or remit (HAMD17< 7 and QIDS-CR rating < 5) with PGx-guided treatment.
Time to response/remission of depressive symptoms. | 8 weeks
  Time to response/remission of depressive symptoms.
Medication change | 8 weeks
  Number of subjects who changed their baseline antidepressant medication regimens.
Health care clinical cost | 8 weeks
  Health care clinical cost (defined by mental health resource utilization).
Report availability | 8 weeks
  Percent of time that the PGx interpretive report is completed and available to the psychiatrist/nurse practitioner prior to seeing the patient.
Medication Choice | 8 weeks
  Proportion of time that the psychiatrist/nurse practitioner prescribed a medication that was recommended by the algorithm.
Physician satisfaction | 8 weeks
  Physician satisfaction with delivery of clinical care (defined by a researcher-developed Likert-based satisfaction survey).
Patient Satisfaction | 8 weeks
  Patient satisfaction with delivery of clinical care (defined by a researcher-developed Likert-based satisfaction survey).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Furmaga, PharmD, Principal Investigator — Pine Rest Mental Health Service